CLINICAL TRIAL: NCT00833547
Title: Effects of Eszopiclone on Sleep-dependent Learning in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Associate Professor of Psychology, Dept. of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Sepracor051
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia
Keywords: sleep; schizophrenia; procedural learning; motor skill
MeSH Terms: conditions — Schizophrenia | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Experimental): 3mg of eszopiclone on two consecutive nights
  Interventions: Drug: eszopiclone
- placebo (Placebo Comparator): placebo capsule that looks identical to eszopiclone capsule on two consecutive nights
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eszopiclone — 3 mg of eszopiclone at bedtime on two consecutive nights
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: placebo — Placebo capsules looking identical to eszopiclone at bedtime on two consecutive nights
  Arms: placebo

SUMMARY:
This study will determine whether eszopiclone will normalize sleep patterns and restore sleep-dependent enhancement of motor skill learning in patients with schizophrenia. The investigators will compare subjects taking a placebo to those taking 3 mg of eszopiclone with regard to: sleep architecture and sleep latency as measured by actigraphy and polysomnography and sleep-dependent motor skill learning.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable outpatients with DSM-IV diagnoses of Schizophrenia

Exclusion Criteria:

* History of neurologic or psychiatric disease other than schizophrenia
* Substance abuse or dependence within the past six months
* Other chronic medical conditions that affect sleep
* Pregnancy/breast feeding
* Hepatic impairment
* Treatment with metabolic inhibitors or inducers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dara S. Manoach, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo capsules that appear identical to eszopiclone capsules on 2 consecutive nights
- Eszopiclone: 3mg of eszopiclone at bedtime for two consecutive nights
Period: Overall Study
Arm/Group | Placebo | Eszopiclone
Started | 13 | 12
Completed | 11 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Eszopiclone: 3mg of eszopiclone at bedtime on 2 consecutive nights
- Placebo: placebo capsule that looks identical to eszopiclone at bedtime on 2 consecutive nights
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10) | 34 (9) | 34 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 10 | 17
Overnight change on finger tapping task [Mean (Standard Deviation); unit: percent change] — The finger tapping task involves pressing four numerically labeled keys on a standard computer keyboard with the fingers of the left hand, repeating a five element sequence (4-1-3-2-4) "as quickly and accurately as possible" for 30s. During both training and test sessions, participants alternated tapping and resting for 30s for a total of 12 tapping trials. The measure was the number of correct sequences per trial. Overnight change was the percent change in correct sequences from the last three training trials to the first three test trials the following morning.
  percent change | 8 (19) | -5 (25) | 2 (23)
sleep spindle density [Mean (Standard Deviation); unit: spindles per minute] — spindles per minute during Stage 2 sleep
  spindles per minute | 1.57 (.56) | 1.08 (.43) | 1.3 (.5)

OUTCOME MEASURES:

1. Primary Outcome: Overnight Change on Finger Tapping Task
Description: The finger tapping task involves pressing four numerically labeled keys on a standard computer keyboard with the fingers of the left hand, repeating a five element sequence (4-1-3-2-4) "as quickly and accurately as possible" for 30s. During both training and test sessions, participants alternated tapping and resting for 30s for a total of 12 tapping trials. The measure was the number of correct sequences per trial. Overnight change was the percent change in correct sequences from the last three training trials to the first three test trials the following morning.
Time Frame: Train on Day 3 and Test on Day 4 of study (experimental nights)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 11
percent change | 21 (25) | 2 (22)

2. Primary Outcome: Sleep Spindle Density During Stage 2 Sleep as Measured by Polysomnography
Description: 2 baseline nights (Days 1 &2); 2 experimental nights (Days 3 &4)
Time Frame: during two nights in an inpatient Clinical Research Center
Measure: Mean (Standard Deviation); unit: spindles per minute during Stage 2 sleep
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 11
spindles per minute during Stage 2 sleep | 1.76 (.55) | 1.07 (.45)

ADVERSE EVENTS:
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No